CLINICAL TRIAL: NCT07021430
Title: Focal Mass Drug Administration for the Prevention of Malaria in Pregnancy: a Pilot Randomized Controlled Trial
Brief Title: Focal Mass Drug Administration for the Prevention of Malaria in Pregnancy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 24-3166; R21AI180728 (NIH)
Record Dates: First submitted 2025-05-14; First posted 2025-06-15 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Malaria Prevention
Keywords: Malaria; Focal mass drug administration; Dihydroartemisinin-piperaquine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A single dose of Dihydroartemisinin Piperaquine (Experimental): A single administration of Dihydroartemisinin Piperaquine as a focal mass drug administration Focal Mass Drug Administration.
  Interventions: Drug: Dihydroartemisinin Piperaquine
- Monthly dose of Dihydroartemisinin Piperaquine (Experimental): Monthly doses of Dihydroartemisinin Piperaquine for household members
  Interventions: Drug: Dihydroartemisinin Piperaquine
- Control (No Intervention): Participants in this arm will receive current standard of care.

INTERVENTIONS:
Drug: Dihydroartemisinin Piperaquine — A single or monthly dose of Dihydroartemisinin Piperaquine based on weight will be taken orally.
  Other Names: Focal Mass Drug Administration
  Arms: A single dose of Dihydroartemisinin Piperaquine; Monthly dose of Dihydroartemisinin Piperaquine

SUMMARY:
The purpose of this study is to demonstrate the feasibility, acceptability, and preliminary effectiveness of a focal mass drug administration program for household members of pregnant women to protect against malaria in pregnancy.

DETAILED DESCRIPTION:
The scientific objective of this pilot study is to demonstrate the feasibility, acceptability, and preliminary effectiveness of a focal mass drug administration program for household members of pregnant women to protect against Malaria in Pregnancy. The hypothesis is that eliminating the parasite reservoir within the household will provide a complementary layer of protection against Malaria in Pregnancy especially when access to care is limited and visits may be delayed or missed.

Aim 1: Determine the feasibility and acceptability of a Focal Mass Drug Administration program with dihydroartemisinin-piperaquine as a novel component of the Malaria in Pregnancy prevention package. The study team will conduct an open-label, randomized pilot study at a primary health center in rural western Uganda. The household members of women presenting to their first antenatal Clinic visit will be randomized 1:1:1: to (i) control (ii) one-time Focal Mass Drug Administration, or (iii) monthly Focal Mass Drug Administration. Using an established implementation framework, the study team will assess process measures such as the proportion of household members reached, willingness to take Dihydroartemisinin Piperaquine, adherence to the course of treatment, and frequency of adverse events.

Aim 2: Estimate the efficacy of Focal Mass Drug Administration to create a "safe zone" in the immediate home environment and ultimately prevent Malaria in Pregnancy. Using the study design outlined in Aim 1, The study team will follow participating pregnant women and associated households through delivery, including longitudinal assessments of P. falciparum infection. As a pilot study, the trial is deliberately not powered for statistical tests of significance, but The study team will measure the incidence of (i) clinical malaria, defined as the presence of typical symptoms (e.g., fever, lethargy) and a positive malaria rapid diagnostic test (Rapid Diagnostic Test), (ii) asymptomatic P. falciparum parasitemia and placental malaria by Polymerase Chain Reaction throughout pregnancy and (iii) the incidence of adverse birth outcomes (e.g., stillbirth, low birth weight). In addition, the study team will measure the prevalence of asymptomatic parasitemia in household members using Rapid Diagnostic Tests at three time points to estimate the effectiveness of Focal Mass Drug Administration at maintaining a parasite-free zone

ELIGIBILITY:
Inclusion Criteria:

* Primary residence (i.e., where a person lives for ≥ 6 months per year) in Kasese District with no plans to change residency in subsequent 6 months
* Able and willing to comply with all study procedures and be available for the duration of the study
* Able and willing to consent to study procedures as documented on informed consent form. For children (age <18 years), parent or guardian must provide consent. Children age ≥8 to 17 years will also be asked to provide written assent.

Each pregnant women will also need to meet additional eligibility criteria:

18 years old or older Presenting to Bugoye Level III Health Center for antenatal care and plan to deliver at Bugoye Level III Health Center (i.e., not planned cesarean section) Gestational age ≤22 weeks Human Immunodeficiency Virus negative

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation:
* Temporary or part-time residence in Kasese District (i.e., where a person lives for < 6 months per year)
* Known plans to move within the next 6 months
* Unable or unwilling to provide consent
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study

In addition, individuals with any of the following will still be eligible to participate (e.g,, complete surveys, provide blood samples) but will not be eligible to receive Dihydroartemisinin Piperaquine if randomized to one of the intervention arms:

* Known arrythmia, QT prolongation, or seizure disorder will not be eligible to receive Dihydroartemisinin Piperaquine
* Use of potentially contraindicated medications outlined in Section 5.6
* Weight <5 kg
* Known allergic reaction to Dihydroartemisinin Piperaquine or other Artemisinin Combination Therapies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percent of eligible household members receiving fMDA | Day 1 to study completion, generally 5 months
  Proportion of eligible household members that receive fMDA intervention according to dosing schedule (i.e., one time or monthly)

SECONDARY OUTCOMES:
Percent of household members enrolled | At enrollment visit (Day 1)
  Proportion of household members who consent to participate
Refusal to receive fMDA | Day 1 to study completion, generally 5 months
  Proportion of eligible household members who decline any fMDA intervention
fMDA Adherence | Day 1 to study completion, generally 5 months
  Proportion of DP blister packs returned with all medication taken (i.e., pill counts)
P. falciparum parasitemia among household members | Day 1 to study completion, generally 5 months
  Prevalence of P. falciparum parasitemia among household members at three time points (enrollment, mid-point, delivery) as measured by malaria rapid diagnostic test
P. falciparum parasitemia among pregnant women | Day 1 to study completion, generally 5 months
  Prevalence of P. falciparum parasitemia as measured by RDT or PCR among women during any point in pregnancy
P. falciparum parasitemia in peripheral and placental blood at delivery | At time of birth/delivery
  Prevalence of P. falciparum parasitemia in peripheral and placental blood at delivery as measured by PCR
Clinical malaria incidence among pregnant women | Day 1 to study completion, generally 5 months
  Incidence of clinical malaria among pregnant women, defined as the presence of acute febrile illness and a positive malaria rapid diagnostic test (RDT)
Maternal anemia | Day 1 to study completion, generally 5 months
  Change in prevalence of maternal anemia, defined as Hemoglobin <11 g/dL among participants
Adverse birth outcomes | Day 1 to study completion, generally 5 months
  Composite of adverse events including spontaneous abortion, premature delivery (<37 weeks gestation), stillbirth, and low birthweight
Co-occurrence of malaria parasitemia in mother and household members | Day 1 to study completion, generally 5 months
  Proportion of RDT+ individuals in each household stratified by parasitemia status of pregnant women at enrollment visit
Number of adverse reactions to DP | Day 1 to study completion, generally 5 months
  Number of dihydroartemisinin-piperaquine administrations that result in vomiting or other known side effects

CONTACTS AND LOCATIONS:
Overall Officials: Ross Boyce, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bugoye Level III Health Center, Kasese, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Requesting investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill.
URL: http://unc.edu